CLINICAL TRIAL: NCT02271282
Title: Pilot Study of Estradiol-Receptor Blockade in Older Men and Women
Brief Title: Estradiol-Receptor Blockade in Older Men and Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Johannes D. Veldhuis, Professor, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 14-004704
Record Dates: First submitted 2014-10-17; First posted 2014-10-22 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Normal Healthy Volunteers
MeSH Terms: interventions — Toremifene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Toremifene/Oral Placebo (Experimental): Oral toremifene will be given once on Day 1 and continue daily x10 days. A single combined IV injection of growth hormone releasing hormone (GHRH)/ghrelin (both doses 0.3mcg/kg) will be given on the overnight visit.
  After at least 3 weeks, subjects will return to receive oral placebo on Day 1 and continue daily x10 days. A single combined IV injection of GHRH/ghrelin (both doses 0.3mcg/kg) will be given on the overnight visit.
  Interventions: Drug: Toremifene; Drug: Placebo; Drug: GHRH/Ghrelin combined Injection
- Oral Placebo/Oral Toremifene (Experimental): Oral placebo will be given once on Day 1 and continue daily x10 days. A single combined IV injection of GHRH/ghrelin (both doses 0.3mcg/kg) will be given on the overnight visit.
  After at least 3 weeks, subjects will return to receive oral toremifene on Day 1 and continue daily x10 days. A single combined IV injection of GHRH/ghrelin (both doses 0.3mcg/kg) will be given on the overnight visit.
  Interventions: Drug: Toremifene; Drug: Placebo; Drug: GHRH/Ghrelin combined Injection

INTERVENTIONS:
Drug: Toremifene
Drug: Placebo
Drug: GHRH/Ghrelin combined Injection

SUMMARY:
Repletion of testosterone (Te) in older men drives GH secretion after its aromatization to estradiol (E2), which acts via the estrogen receptor (ER). Conversely, we postulate that estrogen deprivation in postmenopausal women attenuates growth hormone (GH) secretion and insulin-like growth factor-1 (IGF-I) production, thus favoring development of metabolic syndrome in men treated with toremifene, a new estrogen antagonist used adjunctively in prostatic cancer

DETAILED DESCRIPTION:
Systemic concentrations of Te, E2, GH, IGF-I and insulin growth factor binding protein 3 (IGFBP-3) decline in healthy aging men and women. Relative sex-steroid deprivation accentuates GH and IGF-I depletion, since Te stimulates GH and IGF-I production in older men, hypogonadal males of all ages, and patients undergoing (genotypic female-to-male) gender reassignment. The estrogen-receptor antagonist, tamoxifen, blocks this effect of Te, suggesting involvement of E2 in GH's stimulation at least in young men. E2 alone stimulates GH secretion in young and older women. Because Te is converted to E2 by aromatization in the body, we postulate that E2 is the active moiety in both men and women. Moreover, we hypothesize that the decline of E2 in older men and women contributes to the fall in GH output. These basic concepts will be tested here.

ELIGIBILITY:
Inclusion:

1. 40 healthy women and men (ages 50 to 80 y); women will be post-menopausal (clinically defined by E2 < 50 pg/mL, FSH > 30Iu/L)
2. BMI 18-35 kg/m2
3. community dwelling; and voluntarily consenting

Exclusion:

1. recent use of psychotropic or neuroactive drugs (within five biological half-live);
2. obesity (outside weight range above);
3. Laboratory test results not deemed physician acceptable, viz potassium <3.5 mEq/L, magnesium <1.5 mEq/L, triglycerides > 300, BUN >30 or creatinine > 1.5 mg/dL, liver functions tests twice upper limit of normal, anemia (hemoglobin must meet Blood Bank requirements - Hgb ≥ 12.5 g/dL)
4. drug or alcohol abuse, psychosis, depression, mania or severe anxiety;
5. acute or chronic organ-system disease, including renal failure (creatinine > 1.5 mg/dL)
6. endocrinopathy, other than primary thyroidal failure receiving replacement
7. nightshift work or recent transmeridian travel (exceeding 3 time zones within 7 days of admission),
8. acute weight change (loss or gain of > 2 kg in 6 weeks);
9. allergy to toremifene
10. unwillingness to provide written informed consent.
11. PSA > 4.0 ng/mL in men
12. History or suspicion of prostatic disease (elevated PSA, indeterminate nodule or mass, obstructive uropathy, or breast cancer),
13. Other carcinoma (excluding localized basal cell carcinoma removed or surgically treated with no recurrence).
14. History of thrombotic arterial disease (stroke, TIA, MI, angina) or deep vein thrombophlebitis.
15. History of CHF, cardiac arrhythmias, congenital QT prolongation, and medications used to treat cardiac arrhythmias or other strong CYP3A4 inhibitors.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Summed mass of growth hormone over 10 hours | Participants will be followed for an average of 2 months with growth hormone measurements occuring 10 days after initiating study medication administration.
  Subjects will be given toremifene/placebo on Day 1 to take for 10 days. For one night between Days 8-12, from date of randomization, subjects will undergo a 12-h overnight (2200-1000h) fasting, every 10-min blood sampling. The primary analytical outcome is the summed mass of growth hormone (ie. mean/min/max) secreted in pulses over the first 10h of overnight blood samples. Pulsatile growth hormone is relevant, since sex-steroid hormones and regulatory peptides uniquely control growth hormone secretory-burst mass

SECONDARY OUTCOMES:
Growth hormone responsiveness over last 2h | Participants will be followed for an average of 2 months with growth hormone measurements occuring 10 days after initiating study medication administration
  Subjects will be given toremifene/placebo on Day 1 to take for 10 days. For one night between Days 8-12, from date of randomization, subjects will undergo a 12-h overnight (2200-1000h) fasting, every 10-min blood sampling. The secondary analytical outcome is growth hormone responsiveness over the last 2 hours to bolus GHRH/ghrelin stimulation (ie. mean/min/max).

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Veldhuis, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States